CLINICAL TRIAL: NCT01206244
Title: Diurnal Variation of Tear Meniscus and Tear Osmolarity
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jianhua (Jay) Wang, MD, PhD, Associate Professor, University of Miami
Other Study IDs: UM20100465
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Dry Eye
Keywords: dry eye; tear meniscus; tear osmolarity
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Normal subjects
- Dry eye: clinically diagnosed dry eye with aqueous tear deficiency

SUMMARY:
This study is to determine the diurnal variation of tear meniscus and tear osmolarity in normal subjects and dry eye patients.

DETAILED DESCRIPTION:
This study is to determine the diurnal variation of tear meniscus using OCT and tear osmolarity using Tearlab's osmolarity system in normal subjects and dry eye patients.

ELIGIBILITY:
Inclusion criteria

1. Is at least 18 years old and has full legal capacity to volunteer;
2. Has read and signed the IRB Informed Consent Document;
3. Is willing and able to follow participant instructions;
4. Has clear corneas;
5. Has 20/100 uncorrected visual acuity or better;
6. Is not a hard (or rigid gas permeable) contact lens wearer within the last year;
7. Was a soft contact lens wearer, but stopped wearing at least 1 week ago;
8. Has dry eye according to the study definition of DES (study subjects).

Exclusion criteria

1. Has any systemic disease affecting ocular health except for Sjögren's syndrome;
2. Is using any systemic or topical medications that will affect ocular health except for artificial tears;
3. Has an active ocular disease other than DES, meibomian gland disease or Sjögren's syndrome
4. Has any clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities;
5. Has limbal or bulbar injection or corneal staining that was clinically significant, which are not due to DES;
6. Has worn rigid gas permeable lenses within 1 year;
7. Has had surgery or an eye injury within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects vs. dry eye patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Variations in tear osmolarity and tear meniscus volume in patients with dry eyes and in healthy control subjects over an 8-hr daytime period. | 8 hours
  The mean tear osmolarity of the dry eye patients was 304.0±10.8 mOsm/L, and the mean tear osmolarity of the normal subjects was 298.0±14.2 mOsm/L (P.0.05). Over the course of 8 hrs, the average measured osmolarities of the dry eye group varied by approximately 21.9±13.5 mOsm/L (range, 6-43 mOsm/L), and the average measured tear osmolarities of the normal group varied by approximately 21.0±9.2 mOsm/L (range, 8-35 mOsm/L). At 2:30 PM, the average volume of the tear menisci in the dry eye group was significantly lower than that of the subjects in the normal group (P,0.05). No correlations between the tear meniscus volumes and tear osmolarities of either group were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States